CLINICAL TRIAL: NCT07249931
Title: Efficacy and Safety of Nerivio for the Management of Amplified Musculoskeletal Pain Syndrome in Pediatric Patients: A Nurse Practitioner-Led Pilot Study
Brief Title: Efficacy and Safety of Nerivio for the Management of Amplified Musculoskeletal Pain Syndrome in Pediatric Patients
Acronym: Nerivio
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Health (Other)
Collaborators: Theranica (Industry)
Responsible Party: Principal Investigator, Elizabeth Wong, PNP-PC Pain Management, Principal Investigator, Children's Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nerivio Protocol
Record Dates: First submitted 2025-11-06; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Amplified Musculoskeletal Pain Syndrome (AMPS)
Keywords: Amplified Musculoskeletal Pain Syndrome (AMPS); Pediatrics
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): Patients with AMPS in the control group will use their usual practices to control pain.
  Interventions: Other: Usual Care
- Intervention group (Experimental): Patients in the experimental group will use the Nerivio(R) device once every 48 hours.
  Interventions: Device: Nerivio(R) Device

INTERVENTIONS:
Device: Nerivio(R) Device — Patients will use the Nerivio(R) device once every 48 hours.
  Arms: Intervention group
Other: Usual Care — Patients will use their usual care to treat pain.
  Arms: Control group

SUMMARY:
The goal of this trial is to learn how the Nerivio® device works to treat Amplified Musculoskeletal Pain Syndrome (AMPS) in children ages 8-18. Nerivio® is a wearable device that activates specific nerves in the upper arm. This causes a response from the brain that has been helpful for people who experience migrane headaches. The main questions this study aims to answer are:

* How well does the Nerivio® device help in reducing pain in children with AMPS?
* Does the use of the Nerivio® device help improve quality of life in children with AMPS?
* How satisfied are children and their families with the use of the Nerivio® device for treatment of AMPS?

Researchers will compare the use of the Nerivio® device with usual treatment for AMPS (including pain medications, physical therapy, and other interventions) to see how well the Nerivio® device helps control pain.

Participants will be in one of two groups, decided by:

* Those who are in the "control" group will use their usual practices to control pain.
* Those who are in the "intervention" group will use the Nerivio® device once every other day.

All participants in the "control group" will:

* Complete surveys and answer questions about their pain and how it affects their daily life
* Use their existing methods for pain control.

All participants in the "intervention" group will:

* Complete surveys and answer questions about their pain and how it affects their daily life
* Learn how to work the Nerivio® device and smartphone app.
* Use the Nerivio® device every other day (every 48 hours).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AMPS by a medical provider experienced in pediatric pain management
* Chronic musculoskeletal pain ≥3 months
* Baseline pain intensity of ≥4 on a 0-10/10 Numeric Rating Scale (NRS)
* Able to comprehend and follow instructions for the device use
* Access to compatible smartphone or device to operate the Nerivio app
* Commit to a four-week treatment and data collection period
* Must be age 8 years - 18 years old

Exclusion Criteria:

* Active autoimmune disease.
* Use of implantable electronic medical devices.
* Neurological disorders that impair study participation as determined by the enrolling provider.
* Severe Mood disorders
* Recent change in pain medications or psychotropic medications (within last 4 weeks)
* Currently or plan to be pregnant (Urine or blood HCG testing done upon enrollment)
* Inability to comply with study procedures or use the device as directed

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment | over a four-week intervention period.
  Measure change from baseline in pain scores to reported pain scores after using the Nerivio device for pediatric patients with AMPS.

SECONDARY OUTCOMES:
Frequency of as needed pain medications | 4 weeks
  Evaluate frequency in PRN medications for pain in both the participants using the Nerivio device and those with only the traditional treatment plan.

OTHER OUTCOMES:
Functionality | 4 weeks
  o Examine changes in functional outcomes, including school attendance, physical activity, and quality of life following the use of the device as reported by subjects.
Satisfaction and Adherence of Nerivio Device use | every week for a total of 4 weeks
  Determine patient and caregiver satisfaction and adherence to the Nerivio treatment protocol through a series of question via weekly questionnaire.
Safety and tolerability | 4 weeks
  Evaluate the safety and tolerability of the Nerivio device in the pediatric AMPS population by reviewing any incident reports or complaints from the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No